CLINICAL TRIAL: NCT02952586
Title: A RANDOMIZED DOUBLE-BLIND PHASE 3 STUDY OF AVELUMAB IN COMBINATION WITH STANDARD OF CARE CHEMORADIOTHERAPY (CISPLATIN PLUS DEFINITIVE RADIATION THERAPY) VERSUS STANDARD OF CARE CHEMORADIOTHERAPY IN THE FRONT-LINE TREATMENT OF PATIENTS WITH LOCALLY ADVANCED SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK
Brief Title: Study To Compare Avelumab In Combination With Standard of Care Chemoradiotherapy (SoC CRT) Versus SoC CRT for Definitive Treatment In Patients With Locally Advanced Squamous Cell Carcinoma Of The Head And Neck (JAVELIN HEAD AND NECK 100)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial prematurely terminated as recommended by the E-DMC because the boundary for futility has been crossed.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B9991016; 2016-001456-21 (EudraCT Number); LOCALLY ADVANCED HEAD AND NECK (Other: Alias Study Number)
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — avelumab; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avelumab + SOC Chemoradiation Therapy (Experimental): * Avelumab 10 mg/kg IV: Day 1 of the Lead-in Phase; Days 8, 25, and 39 of the CRT Phase; and Q2W for 12 months during the Maintenance Phase
  * Cisplatin 100 mg/m2 IV: Days 1, 22, and 43 of the CRT Phase
  * Intensity Modulated Radiation Therapy (IMRT) 70 Gy/35 fractions/7 weeks; 1 fraction per day, 5 fractions/week for 7 weeks during the CRT Phase
  Interventions: Drug: Avelumab
- Placebo + SOC CRT (Placebo Comparator): * Placebo IV matching avelumab: Days 1 of the Lead-in Phase; Days 8, 25, and 39 of the CRT Phase; Q2W for 12 months during the Maintenance Phase
  * Cisplatin 100 mg/m2 IV: Days 1, 22, and 43 of the CRT Phase
  * IMRT 70 Gy/35 fractions/7 weeks; 1 fraction per day, 5 fractions/week for 7 weeks during the CRT Phase
  Interventions: Other: Chemoradiation

INTERVENTIONS:
Drug: Avelumab — Avelumab + SOC Chemoradiation
  Arms: Avelumab + SOC Chemoradiation Therapy
Other: Chemoradiation — Cisplatin + Radiation Therapy
  Arms: Placebo + SOC CRT

SUMMARY:
This is a phase 3 randomized, placebo controlled study to evaluate the safety and anti-tumor activity of Avelumab in combination with standard of care chemoradiation (SoC CRT) versus SoC CRT alone in front-line treatment of patients with locally advanced head and neck cancer.

ELIGIBILITY:
INCLUSION CRITERIA

* Histological diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
* HPV negative disease, Stage III, IVa, IVb; non-oropharyngeal HPV positive disease Stage III, IVa, IVb, HPV positive oropharyngeal disease T4 or N2c or N3
* No prior therapy for advanced stage SCCHN; eligible for definitive CRT with curative intent.
* Available tumor samples for submission or willing to undergo further tumor biopsies:
* Age ≥18 years (≥19 in Korea;20 years in Japan and Taiwan).
* ECOG Performance Status 0 or 1
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* Pregnancy test (for patients of childbearing potential) negative at screening

EXCLUSION CRITERIA

* Prior immunotherapy with an anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti CTLA 4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways.
* Major surgery 4 weeks prior to randomization.
* Prior malignancy requiring tumor-directed therapy within the last 2 years prior to enrollment, or concurrent malignancy associated with clinical instability. Exceptions for disease within the 2 years are superficial esophageal cancer (TIS or T1a) fully resected by endoscopy, prostate cancer (Gleason score 6) either curatively treated or deemed to not require treatment, ductal IS carcinoma of the breast that has completed curative treatment, adequately treated basal cell or squamous cell skin cancer.
* Active autoimmune disease
* Any of the following in the 6 months prior to randomization: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
* Active infection requiring systemic therapy.
* Use of immunosuppressive medication at time of randomization
* Prior organ transplantation including allogenic stem-cell transplantation.
* Diagnosis of prior immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Vaccination within 4 weeks prior to randomization.
* Current use of or anticipated need for treatment with other anti-cancer drugs.
* Pregnant female patients, breastfeeding female patients, and male patients able to father children and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study and for at least 6 months after the last dose of cisplatin and 60 days after the last dose of avelumab/placebo (whichever is later).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 697 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (311):
- United States (135):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - The Oncology Institute of Hope and Innovation, Anaheim, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - UCSD Radiation Oncology South Bay, Cancer Treatment Centers, Chula Vista, California
  - City of Hope Corona, Corona, California
  - Compassionate Care Research Group, Inc. at Compassionate Cancer Care Medical Group, Inc., Corona, California
  - The Oncology Institute of Hope and Innovation, Downey, California
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - UC San Diego Medical Center- La Jolla (Thornton Hospital), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - The Oncology Institute of Hope and Innovation, Los Angeles, California
  - Cedars Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Lynwood, California
  - The Oncology Institute of Hope and Innovation, Montebello, California
  - UC Irvine Medical Center, Orange, California
  - Compassionate Care Research Group, Inc. at Compassionate Cancer Care Medical Group, Inc., Riverside, California
  - UC San Diego Medical Center- Hillcrest, San Diego, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - City of Hope South Pasadena, South Pasadena, California
  - The Oncology Institute of Hope and Innovation, Torrance, California
  - The Oncology Institute of Hope and Innovation, West Covina, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Denver CTO/CTRC, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion, Aurora, Colorado
  - University Of Colorado Hospital Cancer Center, Aurora, Colorado
  - Cypress Hematology & Oncology, Denver, Colorado
  - Cypress Hematology and Oncology, Parker, Colorado
  - Sylvester at Coral Gables, Coral Gables, Florida
  - Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Specialist Global LLC, Hialeah, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Hollis Cancer Center, Lakeland, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Sylvester at Plantation, Plantation, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Primary Healthcare Associates, Flossmoor, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Primary Healthcare Associates, Harvey, Illinois
  - Primary Healthcare Associates, Tinley Park, Illinois
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Kansas City VA Radiation Oncology Clinic, Overland Park, Kansas
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University Medical Center, Inc., Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Highlands Cancer Center, Prestonsburg, Kentucky
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Herbert-Herman Cancer Center, Sparrow Hospital, Lansing, Michigan
  - Siteman Cancer Center- St. Peters, City of Saint Peters, Missouri
  - University of Missouri- Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Department of Radiation Oncology Methodist Hospital, Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center-Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center- Bergen, Montvale, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center Westchester, Harrison, New York
  - Bellevue Hospital Center, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Langone Radiology, New York, New York
  - NYU Langone Radiology - Ambulatory Care Center East 41st Street, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center: Breast and Imaging Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Cancer Center- Nassau, Uniondale, New York
  - Oncology Specialists of Charlotte, PA, Charlotte, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center- Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network Cancer Center Pharmacy, Allentown, Pennsylvania
  - Lehigh Valley Health Network-Cedar Crest, Allentown, Pennsylvania
  - Radiation Oncology Cancer Services, Allentown, Pennsylvania
  - Lehigh Valley Health Network-Muhlenberg, Bethlehem, Pennsylvania
  - Precision Cancer Research / Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - PinnacleHealth Cancer Institute, Harrisburg, Pennsylvania
  - PinnacleHealth Cancer Institute, Jacksville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Radiation Oncology, Pittsburgh, Pennsylvania
  - MUSC- Rutledge Tower, Charleston, South Carolina
  - Medical University of South Carolina- Hollings Cancer Center, Charleston, South Carolina
  - MUSC SCTR Research Nexus Clinical Science Building, Charleston, South Carolina
  - MUSC- Ashley River Tower, Charleston, South Carolina
  - MUSC- Radiation Oncology, Charleston, South Carolina
  - MUSC- University Hospital, Charleston, South Carolina
  - GHS Cancer Institute, Easley, South Carolina
  - GHS Cancer Institute, Greenville, South Carolina
  - GHS Cancer Institute, Greer, South Carolina
  - GHS Cancer Institute, Seneca, South Carolina
  - GHS Cancer Institute, Spartanburg, South Carolina
  - The West Clinic, PC dba West Cancer Center, Germantown, Tennessee
  - The West Clinic PC dba West Cancer Center, Memphis, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Texas Oncology El Paso Cancer Treatment Center, El Paso, Texas
  - William Beaumont Army Medical Center, El Paso, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Hospital - TMC, Houston, Texas
  - UTHealth/Memorial Hermann Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Utah Cancer Specialists, Murray, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
- Australia (7):
  - Chris O'Brien Lifehouse Medical Imaging, Camperdown, New South Wales
  - Chris O'Brien Lifehouse Radiation Oncology Department, Camperdown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Northern Sydney Cancer Centre, St Leonards, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
- Ordensklinikum Linz GmbH, Linz, Austria
- Belgium (5):
  - University Hospital Brussels, Brussels
  - Grand Hopital de Charleroi - Site Notre-Dame, Charleroi
  - Centre Hospitalier de Jolimont, Haine-Saint-Paul
  - Site Sainte Elisabeth / CHU UCL Namur, Namur
  - GZA Hospitals Campus Sint Augustinus, Wilrijk
- CHU de Quebec - Universite Laval, Québec, Quebec, Canada
- China (16):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University/Oncology Department, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hai Nan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - Xiangya Hospital Central South University/Oncology Department, Changsha, Hunan
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital/Oncology Department, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
- France (20):
  - Institut de Cancerologie de l'Ouest (ICO) - Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hopital Pellegrin - Service de radiologie et d'imagerie, Bordeaux
  - Hopital Saint-Andre, Bordeaux
  - Cabinet de radiologie Privé - Dr Joseph Mocaer, Brest
  - Clinique Pasteur - CFRO, Brest
  - Hopital Franco-Britannique, Institut d'Oncologie Hauts-de-Seine Nord, Levallois-Perret
  - Institut Regional du Cancer Montpellier - Val d'Aurelle, Montpellier
  - Hopital prive du Confluent S.A.S., Nantes
  - Hopital prive du Confluent S.A.S, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Americain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Institut de Cancerologie de l'Ouest (ICO) - Site Rene Gauducheau, Saint-Herblain
  - Institut de cancerologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss - Radiologie et medecine nucleaire, Strasbourg
  - ICANS - Institut de cancerologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Helios Klinikum Berlin-Buch, Institut fur Rontgendiagnostik, Berlin, BUCH
  - Helios Klinikum Berlin-Buch, Klinik fur Nuklearmedizin, Berlin, BUCH
  - Helios Klinikum Berlin-Buch, Klinik fur Strahlentherapie, Berlin, BUCH
  - Helios Klinikum Berlin-Buch, Berlin, BUCH
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Jena, Jena
  - Universitätsklinikum Regensburg, Regensburg
- Greece (3):
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Athens, Attica
  - Attikon University Hospital, Haidari, Attica
  - Euromedica General Clinic, Thessaloniki
- Hungary (7):
  - Orszagos Onkologiai Intezet, B Belgyogyaszati Osztaly, Budapest
  - Orszagos Onkologiai Intezet, Sugarterapias Osztaly, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Koraz, Onkoradiologiai osztaly, Győr
  - Pecsi Tudomanyegyetem, Klinikai Kozpont, Onkoterapias Intezet, Pécs
  - Szegedi Tudomanyegyetem, Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Ireland (4):
  - St Luke's Radiation Oncology Network, St Luke's Hospital, Dublin
  - St James's Hospital, Dublin
  - St. James's Hospital, Dublin
  - Blackrock Clinic, Dublin
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital, Department of Oncology, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba M.C.Tel-Hashomer, Ramat Gan
- Italy (14):
  - ASST degli Spedali Civili di Brescia, Brescia, BS
  - Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori (I.R.S.T), Meldola, FC
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - Ospedale M. Bufalini, Cesena, Forlì-cesena
  - IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, Forlì-cesena
  - Presidio Ospedaliero Vito Fazzi, Lecce, LE
  - AOU Policlinico Di Modena, Modena, MO
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - UOC Oncologia Medica, AUSL della Romagna -RAVENNA, Lugo, RA
  - IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Ravenna, RA
  - UOC Oncologia Medica, AUSL della Romagna - RAVENNA, Ravenna, RA
  - AULSS 9 - Scaligera Ospedale Mater Salutis, Legnago, VR
  - Istituto Nazionale Tumori IRCCS - Fondazione Pascale, Napoli
  - AUSL - IRCCS and Reggio Emilia, Reggio Emilia
- Japan (15):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Poland (6):
  - Centrum Onkologii im. prof. F. Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii - Instytut im. M. Sklodowskiej - Curie, Klinika Radioterapii i Chemioterapii, Gliwice
  - SPZOZ Ministerstwa Spraw Wewnetrznych i Administracji z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - NZOZ Provita Prolife Centrum Medyczne, Tomaszów Mazowiecki
  - Specjalistyczny Szpital Onkologiczny NU-MED sp. z o.o., Tomaszów Mazowiecki
- Portugal (8):
  - Hospital Pedro Hispano, Matosinhos Municipality, Porto District
  - CUF Porto, Senhora da Hora, Porto District
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Vila Nova de Gaia, Porto District
  - Instituto Portugues de Oncologia de Coimbra Francisco Gentil, E.P.E., Coimbra
  - Centro Hospitalar do Porto, E.P.E.- Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E., Porto
  - Centro Hospitalar São João, E.P.E, Porto
  - Julio Teixeira, Porto
- Russia (6):
  - SBIH "Chelyabinsk Regional Clinical Centre of Oncology and Nuclear Medicine", Chelyabinsk
  - N. N. Blokhin NMRCO, Moscow
  - Budgetary Institution of Healthcare of Omsk Region "Clinical Oncology Dispensary", Omsk
  - FSBI "National Medical Research Center of Oncology n.a. N.N. Petrov", Saint Petersburg
  - SBIH "SPb Clinical Research Centre of Specialized Kinds of Medical Care (Oncology)", Saint Petersburg
  - SBHI YaR "Regional Clinical Oncology Hospital", Yaroslavl
- South Korea (12):
  - Center for Proton Therapy, National Cancer Center, Goyang-si, Gyeonggi-do
  - Center for Specific Organ Cancer, National Cancer Center, Goyang-si, Gyeonggi-do
  - Department of Radiation Oncology, CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Division of Radiation Oncology, Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Division of Radiation Oncology, Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Department of Radiation Oncology, Ulsan University Hospital, Ulsan
  - Ulsan University Hospital, Ulsan
- Spain (16):
  - Institut Catala d'Oncologia Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Institut Catala D'Oncologia de Girona, Girona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Switzerland (12):
  - Klinik fur Radiologie und Nuklearmedizin, Basel, Canton of Basel-City
  - Klinik fur Strahlentherapie und Radioonkologie, Basel, Canton of Basel-City
  - Universitatsspital Basel, Basel, Canton of Basel-City
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Kantonsspital Winterthur, Medizinische Onkologie, Winterthur, Canton of Zurich
  - Kantonsspital Winterthur, Radiologie, Winterthur, Canton of Zurich
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Istituto Oncologico della Svizzera Italiana IOSI, Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Radiologia ORBV, Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Institut fur Klinische Pathologie, Zurich
  - Klinik fur Nuklearmedizin, Zurich
  - Universitatsspital Zurich, Zurich
- Taiwan (7):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital-Linkou Branch, Taoyuan
- United Kingdom (5):
  - NHS Grampian, Aberdeen
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - NHS Lothian, Western General Hospital, Edinburgh
  - Guy's and St. Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lee NY, Ferris RL, Psyrri A, Haddad RI, Tahara M, Bourhis J, Harrington K, Chang PM, Lin JC, Razaq MA, Teixeira MM, Lovey J, Chamois J, Rueda A, Hu C, Dunn LA, Dvorkin MV, De Beukelaer S, Pavlov D, Thurm H, Cohen E. Avelumab plus standard-of-care chemoradiotherapy versus chemoradiotherapy alone in patients with locally advanced squamous cell carcinoma of the head and neck: a randomised, double-blind, placebo-controlled, multicentre, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):450-462. doi: 10.1016/S1470-2045(20)30737-3. PMID 33794205
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 3 sequential treatment phases: Lead-in, CRT, and Maintenance. There were 3 treatments administered in parallel during CRT phase: Avelumab, Cisplatin and IMRT.
Pre-assignment Details: Study had 3 sequential treatment phases: Lead-in, CRT, and Maintenance. There were 3 treatments administered during CRT phase: Avelumab, Cisplatin and IMRT. Reasons for discontinuation of each treatment are summarized separately. 11 participants discontinued all 3 treatments during CRT phase due to death. Two patients discontinued cisplatin due to adverse event and subsequently discontinued avelumab and IMRT due to death.
Groups:
- Avelumab + Standard of Care Chemotherapy (SOC CRT): Participants with locally advanced squamous cell carcinoma of the head and neck (LA SCCHN) were administered with avelumab 10 milligram per kilogram (mg/kg) intravenous (IV) injection on Day 1 of the Lead-in Phase (7 days) and on Days 8, 25 and 39 in CRT phase (63 days). In CRT phase participants also received SOC CRT: cisplatin 100 milligram per square meter (mg/m^2) on Days 1, 22, 43 and intensity-modulated radiation therapy (IMRT) 5 days a week. CRT phase was followed by maintenance phase (12 months) in which participants received avelumab 10 mg/kg IV injection every 2 weeks. All participants were followed for safety 30 days after the last study treatment administration or until the time of initiation of new systemic anticancer treatment. If any concern arose participants were followed up on Day 90 via telephone call thereafter in long term (LT) follow up period every 16 weeks for survival and new systemic anticancer treatment.
- Placebo + SOC CRT: Participants with LA SCCHN were administered with placebo IV injection matched to avelumab on Day 1 of the Lead-in Phase (7 days) and on Days 8, 25 and 39 in CRT phase (63 days). In CRT phase participants also received SOC CRT: cisplatin mg/m^2 on Days 1, 22 and 43 + IMRT 5 days a week. CRT phase was followed by maintenance phase (12 months) in which participants received placebo IV injection every 2 weeks. All participants were followed for safety 30 days after the last study treatment administration or until the time of initiation of new systemic anticancer treatment. If any concern arose participants were followed up on Day 90 via telephone call thereafter in long term follow up period every 16 weeks for survival and new systemic anticancer treatment.
Period: Lead-In Phase (7 Days)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 350 | 347
Safety Analysis Set | 348 | 344
Completed | 345 | 343
Not Completed | 5 | 4
Not completed — Death | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — No Longer Met Eligibility Criteria | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Period: CRT for Avelumab or Placebo (63 Days)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 345 | 340 (All participants who did not withdraw from study after Lead-In phase, entered into CRT phase.)
Completed | 312 | 313
Not Completed | 33 | 27
Not completed — Death | 5 | 8
Not completed — Adverse Event | 12 | 12
Not completed — Physician Decision | 2 | 1
Not completed — Global Deterioration of Health Status | 1 | 0
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 2 | 1
Period: CRT for Cisplatin (63 Days)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 345 (Avelumab, Cisplatin, and IMRT were treatments in CRT phase.) | 340 (Placebo, Cisplatin, and IMRT were treatments in CRT phase.)
Completed | 234 | 236
Not Completed | 111 | 104
Not completed — Death | 3 | 8
Not completed — Adverse Event | 82 | 81
Not completed — Physician Decision | 12 | 10
Not completed — Global Deterioration of Health Status | 1 | 0
Not completed — Withdrawal by Subject | 11 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 1
Period: CRT for IMRT (63 Days)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 345 (Avelumab, Cisplatin, and IMRT were treatments in CRT phase.) | 340 (Placebo, Cisplatin, and IMRT were treatments in CRT phase.)
Completed | 322 | 320
Not Completed | 23 | 20
Not completed — Death | 5 | 8
Not completed — Adverse Event | 5 | 5
Not completed — Global Deterioration of Health Status | 1 | 0
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 0
Period: Maintenance Phase (12 Months)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 291 (All participants who did not withdraw from study after CRT phases, entered into maintenance phase.) | 304 (All participants who did not withdraw from study after CRT phases, entered into maintenance phase.)
Completed | 139 | 177
Not Completed | 152 | 127
Not completed — Death | 17 | 11
Not completed — Progressive disease | 60 | 54
Not completed — Adverse Event | 24 | 21
Not completed — Non-compliance With Study Drug | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Global Deterioration of Health Status | 14 | 5
Not completed — Withdrawal by Subject | 31 | 25
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other | 2 | 1
Not completed — Study Terminated by Sponsor | 1 | 6
Period: Follow-Up Phase (90 Days)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 266 (Participants who did not withdraw study after previous phases, entered in short-term follow up phase.) | 284 (Participants who did not withdraw study after previous phases, entered in short-term follow up phase.)
Completed | 208 | 216
Not Completed | 58 | 68
Not completed — Death | 12 | 10
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 7 | 5
Not completed — Study Terminated by Sponsor | 32 | 50
Period: LT Follow-up (up to 45 Months)
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Started | 247 (Participants who did not withdraw study after previous phases, entered in long-term follow up phase.) | 237 (Participants who did not withdraw study after previous phases, entered in long-term follow up phase.)
Completed | 0 | 0
Not Completed | 247 | 237
Not completed — Death | 51 | 31
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Study Terminated by Sponsor | 187 | 201

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT | Total
Number analyzed (Participants) | 350 | 347 | 697
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.36 (8.56) | 58.88 (9.09) | 59.12 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 290 | 285 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 312 | 312 | 624
  Unknown or Not Reported | 25 | 27 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9 | 10 | 19
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 102 | 86 | 188
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 224 | 229 | 453
  Other | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Modified Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) as Assessed by Investigator
Description: PFS was defined as the time (in months) from the date of randomization to the first documentation of objective progressive disease (PD) per modified RECIST v1.1 as assessed by Investigator or death (due to any cause), whichever occurred first. Analysis was performed using Kaplan Meier method. PD refers to any of following: 1) Locoregional PD confirmed by pathology to verify radiographic changes represent true tumor progression and not radiation effects or non-malignant contrast enhancement. 2) Locoregional clinically detectable progression confirmed by pathology. 3) Surgical removal (salvage) of primary tumor with tumor present on final pathology. 4) Salvage neck dissection greater than (>) 20 weeks after completion of CRT with tumor present on final pathology. 5) Metastatic PD. PFS data was censored on date of last adequate tumor assessment for participants with no PFS event.
Time Frame: From randomization until documented PD or death, censored date, whichever occurred first (up to 37 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 350 | 347
months | NA [16.9 to NA] — Median and upper limit of 95% CI were not reached at the time of primary completion date. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC Chemotherapy (CRT) arm was crossed and the study was terminated. | NA [23.0 to NA] — Median and upper limit of 95% CI were not reached at the time of primary completion date. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated.
Statistical Analysis 1: Comparison: Avelumab + Standard of Care Chemotherapy (SOC CRT) vs Placebo + SOC CRT; Test type: Superiority; p = 0.9199, Log Rank — The treatment arms were compared using a stratified, 1-sided, log rank Test. The three stratification factors were tumor (T) stage (< T4 vs T4), Nodal (N) stage (N0 /N1/N2a/N2b vs N2c/N3), Human papillomavirus (HPV) status (Positive vs Negative); Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.928 to 1.573]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan Meier method.
Time Frame: From randomization to the date of death or censored date, whichever occurred first (up to 37 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 350 | 347
months | NA [NA to NA] — Median and 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated. | NA [NA to NA] — Median and 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated.
Statistical Analysis 1: Comparison: Avelumab + Standard of Care Chemotherapy (SOC CRT) vs Placebo + SOC CRT; Test type: Superiority; p = 0.9372, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.927 to 1.849]

3. Secondary Outcome: Pathologic Complete Response (pCR) Rate in Participants With Salvage Surgery at the Primary Site
Description: pCR was defined as the absence of histologically identifiable residual cancer in any resected specimen. The pCR rate at primary site was estimated by dividing the number of participants with pCR recorded at any visit from randomization until PD per modified RECIST v1.1 or death due to any cause by the number of participants randomized who had salvage surgery at the primary site.
Time Frame: From randomization until PD or death (up to 37 months)
Population: All randomized participants who had salvage surgery at the primary site.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 6 | 7
percentage of participants | 0 [0.0 to 45.9] | 14.3 [0.4 to 57.9]

4. Secondary Outcome: Time to Locoregional Failure Per Modified RECIST v1.1 as Assessed by Investigator
Description: Locoregional failure was defined as the time from the date of randomization to the date of the first documentation of locoregional recurrence or death due to any cause per modified RECIST v1.1 as assessed by Investigator, whichever occurred first. Analysis was performed using Kaplan Meier method.
Time Frame: From the date of randomization to the date of the first documentation of locoregional recurrence or death, whichever occurred first (up to 37 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 350 | 347
months | NA [22.4 to NA] — Median and upper limit of 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated. | NA [25.0 to NA] — Median and upper limit of 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated.
Statistical Analysis 1: Comparison: Avelumab + Standard of Care Chemotherapy (SOC CRT) vs Placebo + SOC CRT; Test type: Superiority; p = 0.9316, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.930 to 1.694]

5. Secondary Outcome: Objective Response Rate (ORR) Per Modified RECIST v1.1 as Assessed by Investigator
Description: Objective response (OR) was defined as a complete response (CR) or partial response (PR) per RECIST v1.1 recorded from randomization until disease progression per modified RECIST v1.1 or death due to any cause. A participant was considered to have achieved an OR if the participant had a CR or PR which did not need to be confirmed at a subsequent assessment. CR for target disease: complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis less than [<] 10 millimeter [mm]). CR for non-target disease: disappearance of all non-target lesions and normalization of tumor marker levels. All lymph nodes must be 'normal' in size (<10 mm short axis) . PR: Greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target measurable lesions. The ORR was estimated by dividing the number of participants with OR (CR or PR) by the number of participants randomized.
Time Frame: From randomization until disease progression or death, whichever occurred first (up to 37 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 350 | 347
percentage of participants | 74.0 [69.1 to 78.5] | 74.9 [70.0 to 79.4]
Statistical Analysis 1: Comparison: Avelumab + Standard of Care Chemotherapy (SOC CRT) vs Placebo + SOC CRT; Test type: Superiority; p = 0.6229, Cochran-Mantel-Haenszel — The treatment arms were compared using a stratified, 1-sided, Cochran-Mantel-Haenszel Test. The 3 stratification factors were tumor stage (< T4 vs T4), Nodal stage (N0 /N1/N2a/N2b vs N2c/N3), HPV status (Positive vs Negative); Odds Ratio (OR) = 0.947, 95% CI 2-sided [0.663 to 1.352]

6. Secondary Outcome: Time to Distant Metastatic Failure Per Modified RECIST v1.1 as Assessed by Investigator
Description: Time to distant metastatic failure or distant metastasis (DM) was defined as the time from the date of randomization to the date of the first documentation of distant metastatic or death due to any cause, whichever occurred first. Distant metastatic disease was defined as new tumor identified at a site distant from the head and neck anatomic region or draining lymph nodes. Analysis was performed using Kaplan Meier method.
Time Frame: From the date of randomization to the date of the first documentation of distant metastatic or death (up to 37 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 350 | 347
months | NA [22.8 to NA] — Median and upper limit of 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated. | NA [NA to NA] — Median and 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated.
Statistical Analysis 1: Comparison: Avelumab + Standard of Care Chemotherapy (SOC CRT) vs Placebo + SOC CRT; Test type: Superiority; p = 0.9061, Log Rank — The treatment arms were compared using a stratified, 1-sided, log rank Test. The three stratification factors were tumor stage (< T4 vs T4), Nodal stage (N0 /N1/N2a/N2b vs N2c/N3), HPV status (Positive vs Negative); Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.909 to 1.624]

7. Secondary Outcome: Duration of Response (DOR) Per Modified RECIST v1.1 as Assessed by Investigator
Description: DOR:time from first documentation of objective tumor response (CR/PR) to first documentation of PD/death due to any cause, whichever occurred first.PR:>=30% decrease under baseline of sum of diameters of all target measurable lesions. CR for target disease:complete disappearance of all target lesions with exception of nodal disease.CR for non-target disease: disappearance of all non-target lesions and normalization of tumor marker levels. PD is any of following:1)Locoregional PD confirmed by pathology to verify radiographic changes denote true tumor progression and not radiation effects or non-malignant contrast enhancement.2)Locoregional clinically detectable progression confirmed by pathology.3)Surgical removal of primary tumor with tumor present on final pathology.4)Salvage neck dissection >20 weeks after completion of CRT with tumor present on final pathology.5)Metastatic PD. DOR data was censored on date of last adequate tumor assessment for participants with no overall response.
Time Frame: From the first documentation of objective tumor response to the first documentation of PD or death or censored date, whichever occurred first (up to 37 months)
Population: Analysis population included all randomized participants who had unconfirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 259 | 260
months | NA [NA to NA] — Median and 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated. | NA [NA to NA] — Median and 95% CI were not reached. At the time of pre-specified interim analysis for the outcome measure, the futility boundaries for the Avelumab +SOC CRT arm was crossed and the study was terminated.

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as Graded by National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. TEAE was defined as event with onset dates occurring during the on-treatment period.
Time Frame: Baseline up to 44 months
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 348 | 344
Participants
  Grade 1 | 10 | 8
  Grade 2 | 30 | 53
  Grade 3 | 224 | 215
  Grade 4 | 59 | 49
  Grade 5 | 22 | 17

9. Secondary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory Parameters
Description: Grade 1 and 3 ranges are: Anemia:Hb:<LLN-10.0,<8.0 g/dL;LC decreased (dec):<LLN-800/mm^3,500-200/mm^3;LC increased (inc):grade 3:>20,000/mm^3:NC dec:<LLN-1500/mm^3;<1000-500/mm^3;PC dec:<LLN-75,000/mm^3;<50,000-25,000/mm^3;WBC dec:<LLN-3000/mm^3;<2000-1000/mm^3;ALT inc:>ULN-3.0*ULN;>5.0-20.0*ULN;ALP & GGT inc:>ULN-2.5*ULN;>5.0-20.0*ULN;AST inc:>ULN-3.0*ULN;>5.0-20.0*ULN;BB inc:>ULN-1.5*ULN;>3.0-10.0*ULN;CH high:>ULN-300 mg/dL;>400-500 mg/dL;CPK inc:>ULN-2.5*ULN;>5*ULN-10*ULN;Hypercalcemia:>ULN-11.5;>12.5-13.5mg/dL;Hyperglycemia:>ULN-160; >250-500mg/dL;Hyperkalemia:>ULN-5.5;>6.0-7.0mmol/L;Hypermagnesemia:>ULN-3.0;>3.0-8.0 mg/dL;Hypernatremia:>ULN-150; >155-160 mmol/L;Hypertriglyceridemia;150-300;>500-1000 mg/dL;Hypoalbuminemia:<LLN-3;<2g/dL;Hypocalcemia:<LLN-8.0;<8.0-7.0mg/dL;Hypokalemia:<LLN-3.0;<3.0-2.5mmol/L;Hypomagnesemia;<LLN-1.2;<0.9-0.7 mg/dL;Hyponatremia:<LLN-130;<130-120mmol/L; Hypophosphatemia:<LLN-2.5;<2.0-1.0mg/dL;lipase & serum amylase inc:>ULN-1.5*ULN;>2.0-5.0*ULN.
Time Frame: Baseline up to 15 months
Population: Safety population include all participants who received at least one dose of study drug. Here "Overall Number of Participants analyzed" signifies number of participants evaluable for this outcome measure and 'Number analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 346 | 340
Participants
  Anemia: New or worsened to grade >=1 | 314 | 311
  Anemia: New or worsened to grade >=3 | 42 | 49
  Lymphocyte Count Decreased: New or worsened to grade >=1 | 336 | 330
  Lymphocyte Count (LC) Decreased: New or worsened to grade >=3 | 279 | 284
  Lymphocyte Count (LC) Increased: New or worsened to grade >=1 | 7 | 7
  Lymphocyte Count Increased: New or worsened to grade >=3 | 0 | 0
  Neutrophil Count (NC) Decreased: New or worsened to grade >=1 | 257 | 237
  Neutrophil Count Decreased: New or worsened to grade >=3 | 120 | 101
  Platelet Count (PC) Decreased : New or worsened to grade >=1 | 157 | 154
  Platelet Count Decreased: New or worsened to grade >=3 | 20 | 7
  White Blood Cell (WBC) Decreased: New or worsened to grade >=1 | 309 | 307
  White Blood Cell Decreased: New or worsened to grade >=3 | 121 | 129
  Alanine aminotransferase (ALT) increased: New or worsened to grade >=1 | 152 | 135
  ALT increased: New or worsened to grade >=3 | 13 | 2
  Alkaline phosphatase increased (ALP): New or worsened to grade >=1 | 72 | 49
  Alkaline phosphatase increased: New or worsened to grade >=3 | 1 | 1
  Aspartate aminotransferase (AST) increased: New or worsened to grade >=1: number analyzed (Participants) | 345 | 340
  Aspartate aminotransferase (AST) increased: New or worsened to grade >=1 | 146 | 111
  Aspartate aminotransferase increased: New or worsened to grade >=3: number analyzed (Participants) | 345 | 340
  Aspartate aminotransferase increased: New or worsened to grade >=3 | 11 | 4
  Blood bilirubin (BB) increased (BB): New or worsened to grade >=1 | 58 | 54
  Blood bilirubin increased: New or worsened to grade >=3 | 9 | 4
  Cholesterol (CH) high: New or worsened to grade >=1: number analyzed (Participants) | 161 | 164
  Cholesterol (CH) high: New or worsened to grade >=1 | 25 | 21
  Cholesterol high: New or worsened to grade >=3: number analyzed (Participants) | 161 | 164
  Cholesterol high: New or worsened to grade >=3 | 0 | 0
  CPK increased: New or worsened to grade >=1: number analyzed (Participants) | 160 | 156
  CPK increased: New or worsened to grade >=1 | 7 | 7
  CPK increased: New or worsened to grade >=3: number analyzed (Participants) | 160 | 156
  CPK increased: New or worsened to grade >=3 | 0 | 1
  Creatinine increased: New or worsened to grade >=1 | 334 | 325
  Creatinine increased: New or worsened to grade >=3 | 36 | 37
  GGT increased: New or worsened to grade >=1: number analyzed (Participants) | 191 | 193
  GGT increased: New or worsened to grade >=1 | 37 | 23
  GGT increased: New or worsened to grade >=3: number analyzed (Participants) | 191 | 193
  GGT increased: New or worsened to grade >=3 | 10 | 5
  Hypercalcemia: New or worsened to grade >=1 | 67 | 59
  Hypercalcemia: New or worsened to grade >=3 | 1 | 5
  Hyperglycemia: New or worsened to grade >=1: number analyzed (Participants) | 345 | 340
  Hyperglycemia: New or worsened to grade >=1 | 144 | 137
  Hyperglycemia: New or worsened to grade >=3: number analyzed (Participants) | 345 | 340
  Hyperglycemia: New or worsened to grade >=3 | 28 | 29
  Hyperkalemia: New or worsened to grade >=1 | 106 | 113
  Hyperkalemia: New or worsened to grade >=3 | 9 | 17
  Hypermagnesemia: New or worsened to grade >=1: number analyzed (Participants) | 346 | 339
  Hypermagnesemia: New or worsened to grade >=1 | 39 | 40
  Hypermagnesemia: New or worsened to grade >=3: number analyzed (Participants) | 346 | 339
  Hypermagnesemia: New or worsened to grade >=3 | 10 | 10
  Hypernatremia: New or worsened to grade >=1 | 22 | 20
  Hypernatremia: New or worsened to grade >=3 | 1 | 0
  Hypertriglyceridemia: New or worsened to grade >=1: number analyzed (Participants) | 162 | 161
  Hypertriglyceridemia: New or worsened to grade >=1 | 35 | 26
  Hypertriglyceridemia: New or worsened to grade >=3: number analyzed (Participants) | 162 | 161
  Hypertriglyceridemia: New or worsened to grade >=3 | 1 | 2
  Hypoalbuminemia: New or worsened to grade >=1 | 195 | 170
  Hypoalbuminemia: New or worsened to grade >=3 | 7 | 5
  Hypocalcemia: New or worsened to grade >=1 | 82 | 88
  Hypocalcemia: New or worsened to grade >=3 | 8 | 14
  Hypoglycemia: New or worsened to grade >=1: number analyzed (Participants) | 345 | 340
  Hypoglycemia: New or worsened to grade >=1 | 56 | 44
  Hypoglycemia: New or worsened to grade >=3: number analyzed (Participants) | 345 | 340
  Hypoglycemia: New or worsened to grade >=3 | 2 | 2
  Hypokalemia: New or worsened to grade >=1 | 140 | 122
  Hypokalemia: New or worsened to grade >=3 | 55 | 49
  Hypomagnesemia: New or worsened to grade >=1: number analyzed (Participants) | 346 | 339
  Hypomagnesemia: New or worsened to grade >=1 | 180 | 158
  Hypomagnesemia: New or worsened to grade >=3: number analyzed (Participants) | 346 | 339
  Hypomagnesemia: New or worsened to grade >=3 | 8 | 12
  Hyponatremia: New or worsened to grade >=1 | 232 | 212
  Hyponatremia: New or worsened to grade >=3 | 74 | 70
  Hypophosphatemia: New or worsened to grade >=1: number analyzed (Participants) | 340 | 339
  Hypophosphatemia: New or worsened to grade >=1 | 108 | 100
  Hypophosphatemia: New or worsened to grade >=3: number analyzed (Participants) | 340 | 339
  Hypophosphatemia: New or worsened to grade >=3 | 21 | 19
  Lipase increased: New or worsened to grade >=1: number analyzed (Participants) | 161 | 154
  Lipase increased: New or worsened to grade >=1 | 19 | 13
  Lipase increased: New or worsened to grade >=3: number analyzed (Participants) | 161 | 154
  Lipase increased: New or worsened to grade >=3 | 11 | 3
  Serum amylase increased: New or worsened to grade >=1: number analyzed (Participants) | 159 | 152
  Serum amylase increased: New or worsened to grade >=1 | 13 | 10
  Serum amylase increased: New or worsened to grade >=3: number analyzed (Participants) | 159 | 152
  Serum amylase increased: New or worsened to grade >=3 | 9 | 5

10. Secondary Outcome: Change From Baseline in Vital Sign - Systolic and Diastolic Blood Pressure
Description: Change from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) measured in sitting position were reported.
Time Frame: Baseline, Lead-in phase: Day1; CRT Phase: Days 1, 8, 22, 25, 39, and 43; Maintenance phase: on Days 1 and 15 in Cycles 1 to 13 and EOT (3 days after the last dose of study drug)
Population: Safety analysis set included all participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified category at each specified time point.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 342 | 336
millimeter of mercury
  DBP: Baseline | 77.8 (10.13) | 78.1 (10.91)
  Lead in Phase: DBP: Change at Day 1: number analyzed (Participants) | 2 | 2
  Lead in Phase: DBP: Change at Day 1 | -3.0 (4.24) | -8.0 (11.31)
  CRT Phase: DBP: Change at Day 1: number analyzed (Participants) | 332 | 322
  CRT Phase: DBP: Change at Day 1 | -1.5 (9.52) | -2.2 (9.91)
  CRT Phase: DBP: Change at Day 8: number analyzed (Participants) | 323 | 315
  CRT Phase: DBP: Change at Day 8 | -3.8 (10.46) | -3.9 (10.99)
  CRT Phase: DBP: Change at Day 22: number analyzed (Participants) | 313 | 309
  CRT Phase: DBP: Change at Day 22 | -4.2 (11.77) | -5.0 (10.95)
  CRT Phase: DBP: Change at Day 25: number analyzed (Participants) | 310 | 306
  CRT Phase: DBP: Change at Day 25 | -3.4 (11.91) | -3.3 (11.44)
  CRT Phase: DBP: Change at Day 39: number analyzed (Participants) | 309 | 302
  CRT Phase: DBP: Change at Day 39 | -5.7 (11.83) | -5.1 (12.14)
  CRT Phase: DBP: Change at Day 43: number analyzed (Participants) | 293 | 283
  CRT Phase: DBP: Change at Day 43 | -5.0 (11.49) | -4.7 (11.76)
  Maintenance Phase: DBP: Change at Cycle1/Day 1: number analyzed (Participants) | 282 | 290
  Maintenance Phase: DBP: Change at Cycle1/Day 1 | -4.8 (11.43) | -4.3 (11.67)
  Maintenance Phase: DBP: Change at Cycle1/Day 15: number analyzed (Participants) | 265 | 279
  Maintenance Phase: DBP: Change at Cycle1/Day 15 | -3.7 (11.78) | -4.0 (10.96)
  Maintenance Phase: DBP: Change at Cycle2/Day 1: number analyzed (Participants) | 266 | 277
  Maintenance Phase: DBP: Change at Cycle2/Day 1 | -3.3 (11.74) | -3.3 (12.31)
  Maintenance Phase: DBP: Change at Cycle2/Day 15: number analyzed (Participants) | 255 | 272
  Maintenance Phase: DBP: Change at Cycle2/Day 15 | -2.7 (11.05) | -2.3 (11.82)
  Maintenance Phase: DBP: Change at Cycle3/Day 1: number analyzed (Participants) | 249 | 262
  Maintenance Phase: DBP: Change at Cycle3/Day 1 | -2.7 (11.37) | -3.6 (11.42)
  Maintenance Phase: DBP: Change at Cycle3/Day 15: number analyzed (Participants) | 234 | 255
  Maintenance Phase: DBP: Change at Cycle3/Day 15 | -2.7 (11.09) | -3.4 (11.10)
  Maintenance Phase: DBP: Change at Cycle4/Day 1: number analyzed (Participants) | 222 | 247
  Maintenance Phase: DBP: Change at Cycle4/Day 1 | -2.2 (12.07) | -3.4 (11.42)
  Maintenance Phase: DBP: Change at Cycle4/Day 15: number analyzed (Participants) | 216 | 240
  Maintenance Phase: DBP: Change at Cycle4/Day 15 | -2.4 (11.38) | -3.3 (11.54)
  Maintenance Phase: DBP: Change at Cycle5/Day 1: number analyzed (Participants) | 210 | 241
  Maintenance Phase: DBP: Change at Cycle5/Day 1 | -2.8 (11.61) | -3.2 (10.88)
  Maintenance Phase: DBP: Change at Cycle5/Day 15: number analyzed (Participants) | 204 | 232
  Maintenance Phase: DBP: Change at Cycle5/Day 15 | -2.5 (11.89) | -3.5 (10.69)
  Maintenance Phase: DBP: Change at Cycle6/Day 1: number analyzed (Participants) | 201 | 226
  Maintenance Phase: DBP: Change at Cycle6/Day 1 | -3.1 (11.21) | -3.8 (11.28)
  Maintenance Phase: DBP: Change at Cycle6/Day 15: number analyzed (Participants) | 198 | 230
  Maintenance Phase: DBP: Change at Cycle6/Day 15 | -3.8 (12.20) | -4.6 (11.43)
  Maintenance Phase: DBP: Change at Cycle7/Day 1: number analyzed (Participants) | 190 | 220
  Maintenance Phase: DBP: Change at Cycle7/Day 1 | -4.1 (11.48) | -4.2 (11.52)
  Maintenance Phase: DBP: Change at Cycle7/Day 15: number analyzed (Participants) | 185 | 214
  Maintenance Phase: DBP: Change at Cycle7/Day 15 | -3.8 (12.05) | -3.8 (10.88)
  Maintenance Phase: DBP: Change at Cycle8/Day 1: number analyzed (Participants) | 173 | 209
  Maintenance Phase: DBP: Change at Cycle8/Day 1 | -2.9 (11.29) | -4.1 (10.95)
  Maintenance Phase: DBP: Change at Cycle8/Day 15: number analyzed (Participants) | 167 | 194
  Maintenance Phase: DBP: Change at Cycle8/Day 15 | -3.4 (11.48) | -4.0 (12.29)
  Maintenance Phase: DBP: Change at Cycle9/Day 1: number analyzed (Participants) | 169 | 198
  Maintenance Phase: DBP: Change at Cycle9/Day 1 | -3.1 (11.78) | -4.2 (10.98)
  Maintenance Phase: DBP: Change at Cycle9/Day 15: number analyzed (Participants) | 162 | 194
  Maintenance Phase: DBP: Change at Cycle9/Day 15 | -2.1 (11.52) | -3.7 (12.07)
  Maintenance Phase: DBP: Change at Cycle10/Day 1: number analyzed (Participants) | 161 | 192
  Maintenance Phase: DBP: Change at Cycle10/Day 1 | -2.2 (11.58) | -3.5 (11.54)
  Maintenance Phase: DBP: Change at Cycle10/Day 15: number analyzed (Participants) | 159 | 191
  Maintenance Phase: DBP: Change at Cycle10/Day 15 | -2.5 (10.90) | -4.4 (11.69)
  Maintenance Phase: DBP: Change at Cycle11/Day 1: number analyzed (Participants) | 146 | 179
  Maintenance Phase: DBP: Change at Cycle11/Day 1 | -2.7 (11.01) | -4.6 (11.23)
  Maintenance Phase: DBP: Change at Cycle11/Day 15: number analyzed (Participants) | 139 | 162
  Maintenance Phase: DBP: Change at Cycle11/Day 15 | -2.9 (10.37) | -3.9 (10.22)
  Maintenance Phase: DBP: Change at Cycle12/Day 1: number analyzed (Participants) | 125 | 156
  Maintenance Phase: DBP: Change at Cycle12/Day 1 | -2.1 (9.51) | -3.5 (11.40)
  Maintenance Phase: DBP: Change at Cycle12/Day 15: number analyzed (Participants) | 115 | 146
  Maintenance Phase: DBP: Change at Cycle12/Day 15 | -3.3 (11.78) | -4.6 (11.19)
  Maintenance Phase: DBP: Change at Cycle13/Day 1: number analyzed (Participants) | 105 | 132
  Maintenance Phase: DBP: Change at Cycle13/Day 1 | -2.0 (9.60) | -3.3 (11.49)
  Maintenance Phase: DBP: Change at Cycle13/Day 15: number analyzed (Participants) | 92 | 118
  Maintenance Phase: DBP: Change at Cycle13/Day 15 | -1.1 (10.22) | -3.8 (11.44)
  DBP: EOT: number analyzed (Participants) | 225 | 210
  DBP: EOT | -2.4 (11.96) | -3.2 (11.17)
  SBP: Baseline | 129.8 (16.42) | 130.5 (17.44)
  Lead in Phase: SBP: Change at Day 1: number analyzed (Participants) | 2 | 2
  Lead in Phase: SBP: Change at Day 1 | -5.5 (2.12) | 12.5 (6.36)
  CRT Phase: SBP: Change at Day 1: number analyzed (Participants) | 332 | 322
  CRT Phase: SBP: Change at Day 1 | -2.5 (15.32) | -3.5 (14.82)
  CRT Phase: SBP: Change at Day 8: number analyzed (Participants) | 323 | 315
  CRT Phase: SBP: Change at Day 8 | -8.3 (17.78) | -8.0 (17.58)
  CRT Phase: SBP: Change at Day 22: number analyzed (Participants) | 313 | 309
  CRT Phase: SBP: Change at Day 22 | -8.9 (18.54) | -8.4 (17.55)
  CRT Phase: SBP: Change at Day 25: number analyzed (Participants) | 310 | 306
  CRT Phase: SBP: Change at Day 25 | -7.9 (19.06) | -5.8 (19.51)
  CRT Phase: SBP: Change at Day 39: number analyzed (Participants) | 309 | 302
  CRT Phase: SBP: Change at Day 39 | -10.6 (20.51) | -10.3 (19.05)
  CRT Phase: SBP: Change at Day 43: number analyzed (Participants) | 293 | 283
  CRT Phase: SBP: Change at Day 43 | -9.6 (18.53) | -9.2 (19.52)
  Maintenance Phase: SBP: Change at Cycle1/Day 1: number analyzed (Participants) | 282 | 290
  Maintenance Phase: SBP: Change at Cycle1/Day 1 | -9.4 (17.97) | -9.4 (20.19)
  Maintenance Phase: SBP: Change at Cycle1/Day 15: number analyzed (Participants) | 265 | 279
  Maintenance Phase: SBP: Change at Cycle1/Day 15 | -9.5 (17.73) | -8.2 (19.58)
  Maintenance Phase: SBP: Change at Cycle2/Day 1: number analyzed (Participants) | 266 | 277
  Maintenance Phase: SBP: Change at Cycle2/Day 1 | -7.0 (18.03) | -7.8 (20.09)
  Maintenance Phase: SBP: Change at /Cycle2/Day 15: number analyzed (Participants) | 255 | 272
  Maintenance Phase: SBP: Change at /Cycle2/Day 15 | -7.9 (18.55) | -6.6 (19.73)
  Maintenance Phase: SBP: Change at Cycle3/Day 1: number analyzed (Participants) | 249 | 262
  Maintenance Phase: SBP: Change at Cycle3/Day 1 | -7.3 (18.93) | -8.5 (18.04)
  Maintenance Phase: SBP: Change at Cycle3/Day 15: number analyzed (Participants) | 234 | 255
  Maintenance Phase: SBP: Change at Cycle3/Day 15 | -8.3 (17.79) | -7.1 (19.90)
  Maintenance Phase: SBP: Change at Cycle4/Day 1: number analyzed (Participants) | 222 | 247
  Maintenance Phase: SBP: Change at Cycle4/Day 1 | -8.4 (18.01) | -8.9 (18.41)
  Maintenance Phase: SBP: Change at Cycle4/Day 15: number analyzed (Participants) | 216 | 240
  Maintenance Phase: SBP: Change at Cycle4/Day 15 | -6.2 (18.20) | -8.2 (19.62)
  Maintenance Phase: SBP: Change at Maintenance/Cycle5/Day 1: number analyzed (Participants) | 210 | 241
  Maintenance Phase: SBP: Change at Maintenance/Cycle5/Day 1 | -7.6 (17.57) | -7.7 (18.69)
  Maintenance Phase: SBP: Change at Cycle5/Day 15: number analyzed (Participants) | 204 | 232
  Maintenance Phase: SBP: Change at Cycle5/Day 15 | -8.4 (18.69) | -7.5 (18.49)
  Maintenance Phase: SBP: Change at Cycle6/Day 1: number analyzed (Participants) | 201 | 226
  Maintenance Phase: SBP: Change at Cycle6/Day 1 | -7.6 (17.67) | -8.3 (18.96)
  Maintenance Phase: SBP: Change at Cycle6/Day 15: number analyzed (Participants) | 198 | 230
  Maintenance Phase: SBP: Change at Cycle6/Day 15 | -7.1 (19.35) | -9.4 (19.56)
  Maintenance Phase: SBP: Change at Cycle7/Day 1: number analyzed (Participants) | 190 | 220
  Maintenance Phase: SBP: Change at Cycle7/Day 1 | -9.0 (18.30) | -8.9 (18.96)
  Maintenance Phase: SBP: Change at Cycle7/Day 15: number analyzed (Participants) | 185 | 214
  Maintenance Phase: SBP: Change at Cycle7/Day 15 | -8.7 (18.10) | -6.8 (18.73)
  Maintenance Phase: SBP: Change at Cycle8/Day 1: number analyzed (Participants) | 173 | 209
  Maintenance Phase: SBP: Change at Cycle8/Day 1 | -6.5 (17.00) | -9.4 (18.65)
  Maintenance Phase: SBP: Change at Cycle8/Day 15: number analyzed (Participants) | 167 | 194
  Maintenance Phase: SBP: Change at Cycle8/Day 15 | -6.8 (16.69) | -7.9 (18.21)
  Maintenance Phase: SBP: Change at Cycle9/Day 1: number analyzed (Participants) | 169 | 198
  Maintenance Phase: SBP: Change at Cycle9/Day 1 | -6.1 (18.49) | -8.1 (18.41)
  Maintenance Phase: SBP: Change at Cycle9/Day 15: number analyzed (Participants) | 162 | 194
  Maintenance Phase: SBP: Change at Cycle9/Day 15 | -6.3 (19.00) | -6.7 (20.28)
  Maintenance Phase: SBP: Change at Cycle10/Day 1: number analyzed (Participants) | 161 | 192
  Maintenance Phase: SBP: Change at Cycle10/Day 1 | -6.1 (19.24) | -7.2 (18.63)
  Maintenance Phase: SBP: Change at Cycle10/Day 15: number analyzed (Participants) | 159 | 191
  Maintenance Phase: SBP: Change at Cycle10/Day 15 | -5.6 (17.07) | -7.7 (18.76)
  Maintenance Phase: SBP: Change at Cycle11/Day 1: number analyzed (Participants) | 146 | 179
  Maintenance Phase: SBP: Change at Cycle11/Day 1 | -6.3 (19.44) | -7.7 (18.86)
  Maintenance Phase: SBP: Change at Cycle11/Day 15: number analyzed (Participants) | 139 | 162
  Maintenance Phase: SBP: Change at Cycle11/Day 15 | -6.3 (18.99) | -7.4 (18.65)
  Maintenance Phase: SBP: Change at Cycle12/Day 1: number analyzed (Participants) | 125 | 156
  Maintenance Phase: SBP: Change at Cycle12/Day 1 | -6.8 (18.25) | -6.1 (20.21)
  Maintenance Phase: SBP: Change at Cycle12/Day 15: number analyzed (Participants) | 115 | 146
  Maintenance Phase: SBP: Change at Cycle12/Day 15 | -7.1 (19.34) | -7.8 (19.12)
  Maintenance Phase: SBP: Change at Cycle13/Day 1: number analyzed (Participants) | 105 | 132
  Maintenance Phase: SBP: Change at Cycle13/Day 1 | -5.8 (20.04) | -6.2 (18.54)
  Maintenance Phase: SBP: Change at Cycle13/Day 15: number analyzed (Participants) | 92 | 118
  Maintenance Phase: SBP: Change at Cycle13/Day 15 | -4.9 (18.82) | -5.6 (19.00)
  SBP: EOT: number analyzed (Participants) | 225 | 210
  SBP: EOT | -7.0 (19.83) | -4.9 (17.97)

11. Secondary Outcome: Change From Baseline in Vital Sign - Pulse Rate
Description: Change from baseline in pulse rate in sitting position in beats per minute was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 342 | 336
beats per minute
  Baseline | 79.9 (13.72) | 86.0 (43.0)
  Lead in Phase: Change at Day 1: number analyzed (Participants) | 2 | 2
  Lead in Phase: Change at Day 1 | -3.5 (0.71) | -8.5 (19.09)
  CRT Phase: Change at Day 1: number analyzed (Participants) | 331 | 322
  CRT Phase: Change at Day 1 | 0.7 (11.70) | 1.3 (10.92)
  CRT Phase: Change at Day 8: number analyzed (Participants) | 323 | 315
  CRT Phase: Change at Day 8 | 1.5 (13.15) | 2.2 (12.42)
  CRT Phase: Change at Day 22: number analyzed (Participants) | 314 | 309
  CRT Phase: Change at Day 22 | 0.5 (13.86) | 2.6 (12.24)
  CRT Phase: Change at Day 25: number analyzed (Participants) | 310 | 306
  CRT Phase: Change at Day 25 | -1.6 (14.87) | -1.2 (13.90)
  CRT Phase: Change at Day 29: number analyzed (Participants) | 10 | 8
  CRT Phase: Change at Day 29 | -11.0 (20.47) | 3.6 (21.29)
  CRT Phase: Change at Day 39: number analyzed (Participants) | 310 | 301
  CRT Phase: Change at Day 39 | 4.0 (15.46) | 4.3 (14.71)
  CRT Phase: Change at Day 43: number analyzed (Participants) | 293 | 283
  CRT Phase: Change at Day 43 | 4.7 (16.82) | 6.1 (14.78)
  Maintenance Phase: Change at Cycle1/Day 1: number analyzed (Participants) | 282 | 291
  Maintenance Phase: Change at Cycle1/Day 1 | 5.1 (16.23) | 7.5 (14.43)
  Maintenance Phase: Change at Cycle1/Day 15: number analyzed (Participants) | 265 | 279
  Maintenance Phase: Change at Cycle1/Day 15 | 3.8 (15.04) | 6.3 (13.65)
  Maintenance Phase: Change at Cycle2/Day 1: number analyzed (Participants) | 266 | 277
  Maintenance Phase: Change at Cycle2/Day 1 | 3.5 (15.30) | 5.9 (14.74)
  Maintenance Phase: Change at Cycle2/Day 15: number analyzed (Participants) | 254 | 272
  Maintenance Phase: Change at Cycle2/Day 15 | 4.1 (15.32) | 4.9 (13.94)
  Maintenance Phase: Change at Cycle3/Day 1: number analyzed (Participants) | 249 | 262
  Maintenance Phase: Change at Cycle3/Day 1 | 3.5 (14.49) | 3.9 (14.37)
  Maintenance Phase: Change at Cycle3/Day 15: number analyzed (Participants) | 234 | 255
  Maintenance Phase: Change at Cycle3/Day 15 | 2.8 (14.73) | 2.8 (14.14)
  Maintenance Phase: Change at Cycle4/Day 1: number analyzed (Participants) | 222 | 247
  Maintenance Phase: Change at Cycle4/Day 1 | 1.8 (14.79) | 3.8 (14.95)
  Maintenance Phase: Change at Cycle4/Day 15: number analyzed (Participants) | 216 | 240
  Maintenance Phase: Change at Cycle4/Day 15 | 1.6 (14.80) | 3.8 (15.02)
  Maintenance Phase: Change at Cycle5/Day 1: number analyzed (Participants) | 210 | 241
  Maintenance Phase: Change at Cycle5/Day 1 | 2.6 (13.88) | 2.9 (14.82)
  Maintenance Phase: Change at Cycle5/Day 15: number analyzed (Participants) | 204 | 232
  Maintenance Phase: Change at Cycle5/Day 15 | 1.6 (15.11) | 3.3 (13.74)
  Maintenance Phase: Change at Cycle6/Day 1: number analyzed (Participants) | 201 | 226
  Maintenance Phase: Change at Cycle6/Day 1 | 1.6 (15.42) | 2.7 (15.72)
  Maintenance Phase: Change at Cycle6/Day 15: number analyzed (Participants) | 198 | 230
  Maintenance Phase: Change at Cycle6/Day 15 | 0.4 (14.04) | 1.4 (13.66)
  Maintenance Phase: Change at Cycle7/Day 1: number analyzed (Participants) | 190 | 220
  Maintenance Phase: Change at Cycle7/Day 1 | -0.1 (14.47) | 2.5 (14.18)
  Maintenance Phase: Change at Cycle7/Day 15: number analyzed (Participants) | 185 | 214
  Maintenance Phase: Change at Cycle7/Day 15 | -0.1 (14.24) | 1.4 (14.33)
  Maintenance Phase: Change at Cycle8/Day 1: number analyzed (Participants) | 173 | 209
  Maintenance Phase: Change at Cycle8/Day 1 | -0.2 (13.84) | 1.0 (13.67)
  Maintenance Phase: Change at Cycle8/Day 15: number analyzed (Participants) | 167 | 194
  Maintenance Phase: Change at Cycle8/Day 15 | -1.5 (14.52) | 1.5 (14.86)
  Maintenance Phase: Change at Cycle9/Day 1: number analyzed (Participants) | 169 | 198
  Maintenance Phase: Change at Cycle9/Day 1 | -1.0 (14.29) | -0.1 (14.06)
  Maintenance Phase: Change at Cycle9/Day 15: number analyzed (Participants) | 162 | 194
  Maintenance Phase: Change at Cycle9/Day 15 | -1.0 (14.20) | 0.2 (14.44)
  Maintenance Phase: Change at Cycle10/Day 1: number analyzed (Participants) | 161 | 192
  Maintenance Phase: Change at Cycle10/Day 1 | -0.9 (13.40) | 0.7 (14.52)
  Maintenance Phase: Change at Cycle10/Day 15: number analyzed (Participants) | 159 | 191
  Maintenance Phase: Change at Cycle10/Day 15 | -0.5 (15.33) | 0.7 (14.66)
  Maintenance Phase: Change at Cycle11/Day 1: number analyzed (Participants) | 145 | 178
  Maintenance Phase: Change at Cycle11/Day 1 | -1.6 (14.57) | 0.2 (14.01)
  Maintenance Phase: Change at Cycle11/Day 15: number analyzed (Participants) | 139 | 162
  Maintenance Phase: Change at Cycle11/Day 15 | -0.2 (13.23) | 0.3 (12.93)
  Maintenance Phase: Change at Cycle12/Day 1: number analyzed (Participants) | 125 | 156
  Maintenance Phase: Change at Cycle12/Day 1 | -0.3 (13.92) | 0.4 (13.67)
  Maintenance Phase: Change at Cycle12/Day 15: number analyzed (Participants) | 115 | 146
  Maintenance Phase: Change at Cycle12/Day 15 | -1.4 (14.92) | -0.5 (12.47)
  Maintenance Phase: Change at Cycle13/Day 1: number analyzed (Participants) | 105 | 132
  Maintenance Phase: Change at Cycle13/Day 1 | -1.4 (14.09) | -0.1 (12.22)
  Maintenance Phase: Change at Cycle13/Day 15: number analyzed (Participants) | 92 | 118
  Maintenance Phase: Change at Cycle13/Day 15 | -1.3 (15.57) | 0.4 (13.24)
  EOT: number analyzed (Participants) | 223 | 210
  EOT | 0.2 (14.73) | 1.9 (14.09)

12. Secondary Outcome: Change From Baseline in the European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) Index Score at CRT Phase and Maintenance Phase
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health status in terms of a single index value or utility score. EQ-5D-5L consisted of two components: a health state profile (descriptive system) and a visual analogue scale (VAS) in which participants rate their overall health status from 0 (worst imaginable) to 100 (best imaginable), where higher scores indicated better health status. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L health status index score range between 0 to 1. Higher score indicated better health status.
Time Frame: Baseline, CRT Phase: Days 1 and 29; Maintenance phase: Cycle 1/Day 1, Cycle 3/Day 1, Cycle 7/Day 1, Cycle 7/Day 15, Cycle 11/Day 1, Cycle 11/Day 15, EOT (3 days after the last dose of study drug)
Population: FAS included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified category at each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 334 | 333
units on a scale
  Baseline | 0.7718 (0.17822) | 0.7615 (0.18517)
  CRT Phase: Change at Day 1: number analyzed (Participants) | 321 | 318
  CRT Phase: Change at Day 1 | -0.0078 (0.13269) | 0.0176 (0.14066)
  CRT Phase: Change at Day 29: number analyzed (Participants) | 293 | 276
  CRT Phase: Change at Day 29 | -0.0915 (0.22053) | -0.0487 (0.19175)
  Maintenance Phase: Change at Cycle1/Day1: number analyzed (Participants) | 272 | 279
  Maintenance Phase: Change at Cycle1/Day1 | -0.0749 (0.22126) | -0.0519 (0.17253)
  Maintenance Phase: Change at Cycle3/Day1: number analyzed (Participants) | 239 | 243
  Maintenance Phase: Change at Cycle3/Day1 | -0.0203 (0.21340) | -0.0160 (0.18179)
  Maintenance Phase: Change at Cycle7/Day1: number analyzed (Participants) | 95 | 113
  Maintenance Phase: Change at Cycle7/Day1 | 0.0088 (0.16690) | 0.0140 (0.16240)
  Maintenance Phase: Change at Cycle7/Day15: number analyzed (Participants) | 59 | 79
  Maintenance Phase: Change at Cycle7/Day15 | 0.0552 (0.18544) | 0.0472 (0.17990)
  Maintenance Phase: Change at Cycle11/Day1: number analyzed (Participants) | 90 | 111
  Maintenance Phase: Change at Cycle11/Day1 | 0.0376 (0.21078) | 0.0792 (0.19287)
  Maintenance Phase: Change at Cycle11/Day15: number analyzed (Participants) | 36 | 40
  Maintenance Phase: Change at Cycle11/Day15 | 0.0673 (0.17227) | 0.0389 (0.18732)
  Maintenance Phase: Change at End of treatment: number analyzed (Participants) | 184 | 187
  Maintenance Phase: Change at End of treatment | -0.0051 (0.24528) | 0.0074 (0.24874)

13. Secondary Outcome: Change From Baseline in the European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) VAS Score at CRT Phase and Maintenance Phase
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health status in terms of a single index value or utility score. EQ-5D-5L consisted of two components: a health state profile (descriptive system) and a visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L health status index score range between 0 to 1. Higher score indicated worse health status. In VAS participants rate their overall health status from 0 (worst imaginable) to 100 (best imaginable), where higher scores indicated better health status.
Time Frame: as for outcome 12
Population: FAS included all randomized participants. FAS included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified category at each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 333 | 330
units on a scale
  Baseline | 75.8 (18.20) | 74.9 (18.24)
  CRT Phase: Change at Day 1: number analyzed (Participants) | 317 | 314
  CRT Phase: Change at Day 1 | -1.1 (13.49) | -1.4 (11.39)
  CRT Phase: Change at Day 29: number analyzed (Participants) | 291 | 271
  CRT Phase: Change at Day 29 | -10.9 (19.94) | -9.2 (18.70)
  Maintenance Phase: Change at Cycle1/Day1: number analyzed (Participants) | 272 | 277
  Maintenance Phase: Change at Cycle1/Day1 | -7.7 (19.05) | -6.2 (18.67)
  Maintenance Phase: Change at Cycle3/Day1: number analyzed (Participants) | 240 | 236
  Maintenance Phase: Change at Cycle3/Day1 | -1.8 (18.00) | -0.7 (16.14)
  Maintenance Phase: Change at Cycle7/Day1: number analyzed (Participants) | 95 | 113
  Maintenance Phase: Change at Cycle7/Day1 | -0.6 (14.91) | 8.6 (81.42)
  Maintenance Phase: Change at Cycle7/Day15: number analyzed (Participants) | 59 | 78
  Maintenance Phase: Change at Cycle7/Day15 | 4.8 (18.52) | 3.1 (19.28)
  Maintenance Phase: Change at Cycle11/Day1: number analyzed (Participants) | 89 | 108
  Maintenance Phase: Change at Cycle11/Day1 | 0.3 (17.60) | 4.3 (16.10)
  Maintenance Phase: Change at Cycle11/Day15: number analyzed (Participants) | 37 | 40
  Maintenance Phase: Change at Cycle11/Day15 | 10.1 (24.69) | 2.4 (18.20)
  Maintenance Phase: Change at End of treatment: number analyzed (Participants) | 183 | 184
  Maintenance Phase: Change at End of treatment | -1.9 (22.55) | 0.7 (19.28)

14. Secondary Outcome: Change From Baseline in National Cancer Comprehensive Network Head and Neck Symptom Index-22 Item Scores (NCCN FHNSI-22) at CRT Phase and Maintenance Phase
Description: The NCCN FHNSI-22 questionnaire measured disease symptoms, treatment side effects and overall quality of life in participants with head and neck cancer. The questionnaire contained 22 items with 5-point Likert scales ranging from 0 to 4 as follows: 'not at all = 0', a little bit = 1, somewhat = 2, quite a bit = 3 and very much = 4. Total score ranged from 0 to 88 where, higher scores represented better symptomatology, quality of life or functioning.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 333 | 331
units on a scale
  Baseline | 60.56 (13.731) | 61.05 (13.155)
  CRT Phase: Change at Day 1: number analyzed (Participants) | 318 | 317
  CRT Phase: Change at Day 1 | -0.59 (8.719) | -0.14 (9.136)
  CRT Phase: Change at Day 29: number analyzed (Participants) | 294 | 275
  CRT Phase: Change at Day 29 | -14.34 (16.847) | -14.56 (15.470)
  CRT Phase: Change at Cycle1/Day1: number analyzed (Participants) | 272 | 281
  CRT Phase: Change at Cycle1/Day1 | -11.33 (16.054) | -12.08 (14.950)
  CRT Phase: Change at Cycle3/Day1: number analyzed (Participants) | 241 | 241
  CRT Phase: Change at Cycle3/Day1 | -3.81 (14.017) | -2.26 (13.625)
  CRT Phase: Change at Cycle7/Day1: number analyzed (Participants) | 96 | 113
  CRT Phase: Change at Cycle7/Day1 | -0.86 (12.503) | -0.51 (14.585)
  CRT Phase: Change at Cycle7/Day15: number analyzed (Participants) | 61 | 78
  CRT Phase: Change at Cycle7/Day15 | 3.96 (14.035) | 0.92 (14.454)
  CRT Phase: Change at Cycle11/Day1: number analyzed (Participants) | 88 | 110
  CRT Phase: Change at Cycle11/Day1 | 2.68 (13.367) | 4.90 (14.207)
  CRT Phase: Change at Cycle11/Day15: number analyzed (Participants) | 37 | 40
  CRT Phase: Change at Cycle11/Day15 | 3.96 (14.322) | 3.37 (12.689)
  CRT Phase: Change at End of treatment: number analyzed (Participants) | 184 | 187
  CRT Phase: Change at End of treatment | -2.35 (17.428) | 0.79 (16.509)

15. Secondary Outcome: Programmed Death Receptor-1 Ligand-1 (PD-L1) Biomarker Expression in Tumor Tissue as Assessed by Immunohistochemistry (IHC)
Description: PD-L1 biomarker expression in tumor tissue as assessed by IHC in the form of positive immune cells and tumor staining cells.
Time Frame: Baseline (prior to first dose)
Population: Biomarker analysis set was a subset of the safety analysis set included participants who had at least one screening biomarker assessment. Here' 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: % of PD-L1+ cells
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 299 | 307
% of PD-L1+ cells
  Positive Immune Cells | 7.4 (7.06) | 8.3 (8.47)
  Tumor Staining Cells | 12.7 (24.90) | 18.3 (31.12)

16. Secondary Outcome: Mean Percentage (%) of Total Tumor Area Occupied by Cluster of Differentiation 8 (CD8+) Cells
Description: Description: CD8+ cells are the type of T-lymphocytes. Mean percentage of total tumor area occupied by CD8+ Cells has been reported. Area was measured in millimeter square (mm^2).
Time Frame: Baseline (prior to first dose)
Population: Biomarker analysis set included all participants who had received at least one dose of study drug and who had at least one screening biomarker assessment. Here, 'Overall number of participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: % of tumor area occupied by CD8+ cells
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 289 | 294
% of tumor area occupied by CD8+ cells | 4.9 (6.03) | 5.8 (6.55)

17. Secondary Outcome: Percentage of Participants With Positive and Negative Pathology of Neck Dissection
Description: Percentage of participants with positive and negative pathology of neck dissection were reported. Positive pathology included live tumor cells present or 10% or greater vital tumor tissues. Negative pathology included no live tumor cells present, complete tumor regression, no evidence of vital tumor tissues, less than 10% vital tumor tissue, or not consistent with disease under study.
Time Frame: From randomization until PD as per investigator assessment (up to 37 months)
Population: Analysis population included all participants who had received at least one dose of study drug and who had salvage neck dissection.
Measure: Number; unit: percentage of participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 14 | 15
percentage of participants
  Negative Pathology | 7.14 | 26.70
  Positive pathology | 71.43 | 40.00
  Pathology not reported | 21.43 | 33.30

18. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Avelumab
Description: Maximum observed plasma concentration (Cmax) of Avelumab is reported.
Time Frame: Pre-dose and end of infusion on Day 1 of lead-in phase, Days 8, 25 of CRT phase, Day 1 of Cycle 1 and 2 (each cycle 28 days)
Population: PK concentration analysis was a subset of the safety analysis set and included participants who had at least one post-dose concentration measurement above the lower limit of quantitation (LLQ) for avelumab or cisplatin. Here' 'overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Groups:
- Avelumab + Standard of Care Chemotherapy (SOC CRT): Participants with LA SCCHN were administered with avelumab 10 mg/kg intravenous (IV) injection on Day 1 of the Lead-in Phase (7 days) and on Days 8, 25 and 39 in CRT phase (63 days). In CRT phase participants also received SOC CRT: cisplatin 100 mg/m^2 on Days 1, 22, 43 and IMRT 5 days a week. CRT phase was followed by maintenance phase (12 months) in which participants received avelumab 10 mg/kg IV injection every 2 weeks. All participants were followed for safety 30 days after the last study treatment administration or until the time of initiation of new systemic anticancer treatment. If any concern arose participants were followed up on Day 90 via telephone call thereafter in long term (LT) follow up period every 16 weeks for survival and new systemic anticancer treatment.
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT)
Number analyzed (Participants) | 236
microgram per milliliter
  Lead-in/Day 1 | 203.6 (31)
  CRT/Day 8: number analyzed (Participants) | 207
  CRT/Day 8 | 190.9 (66)
  CRT/Day 25: number analyzed (Participants) | 189
  CRT/Day 25 | 162.4 (114)
  Cycle 1 Day 1: number analyzed (Participants) | 152
  Cycle 1 Day 1 | 142 (117)
  Cycle 2 Day 1: number analyzed (Participants) | 128
  Cycle 2 Day 1 | 154.9 (97)

19. Secondary Outcome: Predose Plasma Concentration (Ctrough) of Avelumab
Description: Ctrough refers to plasma concentration of Avelumab observed just before treatment administration.
Time Frame: Pre-dose on Day 1 of lead-in phase, Days 8, 25 of CRT phase, Day 1 of Cycle 1, 2, 5, 8, 11 (each cycle 28 days)
Population: PK concentration analysis was a subset of the safety analysis set and included participants who had at least one post-dose concentration measurement above the LLQ for avelumab or cisplatin. Here' 'overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT)
Number analyzed (Participants) | 267
microgram per milliliter
  Lead-in/Day 1: number analyzed (Participants) | 263
  Lead-in/Day 1 | 2.988 (1590)
  CRT/Day 8 | 11.9 (63)
  CRT/Day 25: number analyzed (Participants) | 251
  CRT/Day 25 | 6.284 (138)
  Cycle 1/Day 1: number analyzed (Participants) | 183
  Cycle 1/Day 1 | 2.354 (131)
  Cycle 2/Day 1: number analyzed (Participants) | 198
  Cycle 2/Day 1 | 17.56 (70)
  Cycle 5/Day 1: number analyzed (Participants) | 147
  Cycle 5/Day 1 | 24.35 (66)
  Cycle 8/Day 1: number analyzed (Participants) | 125
  Cycle 8/Day 1 | 29.59 (69)
  Cycle 11/Day 1: number analyzed (Participants) | 113
  Cycle 11/Day 1 | 30.85 (79)

20. Secondary Outcome: Dose Normalized Maximum Plasma Concentration (Cmax [dn]) of Total and Free Cisplastin
Description: Dose normalized (dn) Cmax was calculated by dividing Cmax by the exact dose of total and free Cisplastin (in mg) administered to a participant.
Time Frame: Pre-dose, mid-infusion, end of infusion, 3, 4, and 24 hours post dose on Day 1 of CRT phase
Population: PK concentration analysis was a subset of the safety analysis set and included participants who had at least one post-dose concentration measurement above the LLQ for avelumab or cisplatin. Here' 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter per milligram
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 12 | 23
nanogram per milliliter per milligram
  Total Cisplastin | 26.23 (36) | 25.33 (26)
  Free Cisplastin | 11.84 (29) | 7.286 (96)

21. Secondary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast[dn]) of Total and Free Cisplatin
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast). AUClast (dn) was calculated by dividing AUClast by the exact dose of cisplastin (in mg) administered to a participant.
Time Frame: Pre-dose, mid-infusion, end of infusion, 3, 4, and 24 hours post dose on Day 1 of CRT phase
Population: PK concentration analysis was a subset of the safety analysis set and included participants who had at least one post-dose concentration measurement above the LLQ for avelumab or cisplatin. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter/milligram
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 10 | 20
nanogram*hour/milliliter/milligram
  Total Cisplatin | 299.1 (30) | 332.7 (17)
  Free Cisplatin | 36.53 (51) | 29.08 (49)

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Total and Free Cisplatin
Description: Maximum observed plasma concentration (Cmax) of total and free Cisplatin is reported.
Time Frame: Pre-dose, mid-infusion, end of infusion, 3, 4, and 24 hours post dose on Day 1 of CRT phase
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 12 | 23
nanogram per milliliter
  Total Cisplatin | 3781 (44) | 4001 (34)
  Free Cisplatin | 1710 (53) | 1151 (109)

23. Secondary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Total and Free Cisplatin
Description: Time to reach maximum observed plasma concentration (Tmax) of total and free Cisplatin.
Time Frame: Pre-dose, mid-infusion, end of infusion, 3, 4, and 24 hours post dose on Day 1 of CRT phase
Population: PK concentration analysis was a subset of the safety analysis set and included participants who had at least one post-dose concentration measurement above the lower limit of quantitation (LLQ) for avelumab or cisplatin. Here' 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 12 | 23
hour
  Total Cisplatin | 1.000 [0.500 to 2.40] | 1.170 [0.983 to 24.0]
  Free Cisplatin | 1.000 [0.500 to 1.17] | 1.000 [0.500 to 2.12]

24. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Avelumab by Never and Ever Positive Status
Description: ADA never-positive was defined as no positive ADA results at any time point; ADA-negative participants (titer less than< cut point) and ADA ever-positive was defined as at least one positive ADA result at any time point; ADA-positive participants (titer greater than or equal to cut point)
Time Frame: pre-dose on Day 1 up to 30 Days after the end of treatment
Population: Immunogenicity analysis set was a subset of the safety analysis set which included participants who had at least 1 ADA/nAb sample collected for avelumab in Avelumab + Standard of Care Chemotherapy (SOC CRT) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT)
Number analyzed (Participants) | 331
Participants
  ADA never-positive | 277
  ADA ever-positive | 54

25. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Avelumab by Never and Ever Positive Status
Time Frame: Day 1 of lead-in phase and on Days 8 and 25 of CRT phase
Population: Since the study was terminated, sponsor decided not to collect data for nAb, hence not reported.
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 44 months
Description: Same event may appear as AE, serious AE, here distinct events are presented. Event may be serious in 1 participant and non-serious in another or 1 participant may have experienced both serious, non-serious event. Safety analysis set evaluated. Discontinuation during CRT phase due to death is the discontinuation reason for treatments received at the time of event in the treatment disposition summary.All deaths reported as reason of discontinuation at any phase are included in all-cause mortality.
Arm/Group | Avelumab + Standard of Care Chemotherapy (SOC CRT) | Placebo + SOC CRT
All-Cause Mortality (participants affected / at risk) | 86/348 | 62/344
Serious Adverse Events (participants affected / at risk) | 184/348 | 177/344
Other Adverse Events (participants affected / at risk) | 344/348 | 340/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Standard of Care Chemotherapy (SOC CRT) (N=348) | Placebo + SOC CRT (N=344)
Anaemia (Blood and lymphatic system disorders) | 8 | 12
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 3
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Pterygium (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 15 | 13
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 2
Mouth swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 9
Odynophagia (Gastrointestinal disorders) | 3 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 4
Tongue haemorrhage (Gastrointestinal disorders) | 2 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 13
Asthenia (General disorders) | 2 | 6
Chest pain (General disorders) | 2 | 1
Chills (General disorders) | 2 | 0
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 2 | 1
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 1 | 6
Hyperpyrexia (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 2
Hypothermia (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 5 | 6
Pain (General disorders) | 0 | 2
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 12 | 3
Sudden death (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 2
Device related infection (Infections and infestations) | 2 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis candida (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 0
Epididymitis (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 3
Infectious pleural effusion (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Oral infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 25 | 20
Pneumonia bacterial (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Stoma site abscess (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Vascular device infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pancreatic injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 2
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 3 | 2
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 7 | 6
C-reactive protein increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 6 | 3
White blood cell count decreased (Investigations) | 0 | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 9 | 15
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Brain hypoxia (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Subacute combined cord degeneration (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Device dislocation (Product Issues) | 1 | 3
Device malfunction (Product Issues) | 1 | 0
Embedded device (Product Issues) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Delirium (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 12 | 11
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 4
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy (Surgical and medical procedures) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 4
Lymphorrhoea (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Vascular rupture (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Standard of Care Chemotherapy (SOC CRT) (N=348) | Placebo + SOC CRT (N=344)
Anaemia (Blood and lymphatic system disorders) | 206 | 192
Leukopenia (Blood and lymphatic system disorders) | 64 | 46
Lymphopenia (Blood and lymphatic system disorders) | 33 | 27
Neutropenia (Blood and lymphatic system disorders) | 102 | 98
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 41
Ear pain (Ear and labyrinth disorders) | 23 | 12
Hypoacusis (Ear and labyrinth disorders) | 29 | 30
Tinnitus (Ear and labyrinth disorders) | 59 | 66
Hyperthyroidism (Endocrine disorders) | 24 | 7
Hypothyroidism (Endocrine disorders) | 51 | 45
Abdominal pain (Gastrointestinal disorders) | 11 | 20
Abdominal pain upper (Gastrointestinal disorders) | 14 | 18
Constipation (Gastrointestinal disorders) | 178 | 155
Diarrhoea (Gastrointestinal disorders) | 83 | 66
Dry mouth (Gastrointestinal disorders) | 151 | 158
Dyspepsia (Gastrointestinal disorders) | 23 | 21
Dysphagia (Gastrointestinal disorders) | 143 | 152
Nausea (Gastrointestinal disorders) | 210 | 199
Odynophagia (Gastrointestinal disorders) | 62 | 48
Oral pain (Gastrointestinal disorders) | 39 | 43
Stomatitis (Gastrointestinal disorders) | 92 | 96
Vomiting (Gastrointestinal disorders) | 112 | 121
Asthenia (General disorders) | 63 | 58
Chills (General disorders) | 39 | 7
Fatigue (General disorders) | 116 | 127
Localised oedema (General disorders) | 22 | 20
Malaise (General disorders) | 20 | 23
Mucosal inflammation (General disorders) | 146 | 131
Oedema peripheral (General disorders) | 19 | 16
Pain (General disorders) | 23 | 28
Pyrexia (General disorders) | 87 | 45
Oral candidiasis (Infections and infestations) | 25 | 31
Pneumonia (Infections and infestations) | 36 | 25
Upper respiratory tract infection (Infections and infestations) | 24 | 21
Infusion related reaction (Injury, poisoning and procedural complications) | 24 | 6
Radiation skin injury (Injury, poisoning and procedural complications) | 135 | 136
Alanine aminotransferase increased (Investigations) | 56 | 30
Amylase increased (Investigations) | 22 | 10
Aspartate aminotransferase increased (Investigations) | 55 | 26
Blood alkaline phosphatase increased (Investigations) | 22 | 9
Blood creatinine increased (Investigations) | 88 | 73
Blood urea increased (Investigations) | 18 | 17
Gamma-glutamyltransferase increased (Investigations) | 23 | 15
Lymphocyte count decreased (Investigations) | 40 | 42
Neutrophil count decreased (Investigations) | 64 | 60
Platelet count decreased (Investigations) | 40 | 33
Weight decreased (Investigations) | 157 | 171
White blood cell count decreased (Investigations) | 69 | 64
Decreased appetite (Metabolism and nutrition disorders) | 128 | 124
Dehydration (Metabolism and nutrition disorders) | 31 | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 33
Hyperkalaemia (Metabolism and nutrition disorders) | 34 | 32
Hypoalbuminaemia (Metabolism and nutrition disorders) | 42 | 36
Hypocalcaemia (Metabolism and nutrition disorders) | 29 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 87 | 71
Hypomagnesaemia (Metabolism and nutrition disorders) | 93 | 84
Hyponatraemia (Metabolism and nutrition disorders) | 83 | 68
Hypophosphataemia (Metabolism and nutrition disorders) | 23 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 30 | 25
Dizziness (Nervous system disorders) | 41 | 33
Dysgeusia (Nervous system disorders) | 106 | 119
Headache (Nervous system disorders) | 44 | 41
Neuropathy peripheral (Nervous system disorders) | 11 | 28
Anxiety (Psychiatric disorders) | 26 | 34
Depression (Psychiatric disorders) | 10 | 18
Insomnia (Psychiatric disorders) | 57 | 47
Acute kidney injury (Renal and urinary disorders) | 18 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 63
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 51 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 33
Hiccups (Respiratory, thoracic and mediastinal disorders) | 26 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 75 | 92
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 24 | 23
Productive cough (Respiratory, thoracic and mediastinal disorders) | 40 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 20
Dermatitis (Skin and subcutaneous tissue disorders) | 52 | 42
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 24
Erythema (Skin and subcutaneous tissue disorders) | 24 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 24
Rash (Skin and subcutaneous tissue disorders) | 43 | 36
Hypertension (Vascular disorders) | 32 | 28
Hypotension (Vascular disorders) | 22 | 14
Lymphoedema (Vascular disorders) | 18 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT02952586/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02952586/SAP_001.pdf